CLINICAL TRIAL: NCT05728320
Title: Analysis of Glycemic Patterns of Patients Undergoing Bariatric Surgery and Assessment of Risk Factors Capable of Predicting High Glycemic Variability and Unnoticed Hypoglycemia
Brief Title: Glycemic Patterns After Bariatric Surgery and High Glycemic Variability and Hypoglycemia Unawareness Risk Factors
Status: Recruiting | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Principal Investigator, Rio de Janeiro State University
Other Study IDs: Bariglivar
Record Dates: First submitted 2023-01-03; First posted 2023-02-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery
Keywords: Hypoglycemia; Cognition; Glycemic variability; Bariatric surgery
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Gastric bypass: Subjects submitted to gastric bypass
  Interventions: Device: Glucose monitoring with flash glucose monitor
- Sleeve gastrectomy: Subjects submitted to sleeve gastrectomy
  Interventions: Device: Glucose monitoring with flash glucose monitor
- Normal control subjects: Subjects not submitted to bariatric surgery with IMC < 25
  Interventions: Device: Glucose monitoring with flash glucose monitor
- Obese control subjects: Subjects not submitted to bariatric surgery with IMC > 30
  Interventions: Device: Glucose monitoring with flash glucose monitor

INTERVENTIONS:
Device: Glucose monitoring with flash glucose monitor — All groups will be monitorized with a flash glucose monitor and compared after 7-14 days.

SUMMARY:
To study the glycemic patterns of patients undergoing bariatric surgery and what are the risk factors capable of predicting episodes of unnoticed hypoglycemia and high glycemic variability, evaluating patients who underwent reduction gastroplasty with Roux-en-Y reconstruction (GRYR) and sleeve gastrectomy (SG)

DETAILED DESCRIPTION:
To study the glycemic patterns of patients undergoing bariatric surgery and what are the risk factors capable of predicting episodes of unnoticed hypoglycemia and high glycemic variability, evaluating patients who underwent reduction gastroplasty with Roux-en-Y reconstruction (GRYR) and sleeve gastrectomy (SG). Methods: Patients of both sexes, aged 18-60 years, submitted to GRYR and SG, for at least one year, under medical follow-up at the Multiuser Clinical Research Center (CePeM). Patients using hypoglycemic drugs (biguanides, sulfonylureas, glinides, acarbose, GLP-1 analogues, SGLT-2 inhibitors, DPP-IV inhibitors and insulin) and hyperglycemic drugs (corticosteroids, high-dose thiazide diuretics, beta-blockers, diazoxide and octreotide), very restrictive diets (intermittent fasting or ketogenic diet), pregnant women, kidney, heart and/or liver failure, history of neurological disorder, visual or hearing impairment, being treated for alcohol or drug abuse, severe psychiatric disorders (schizophrenia, bipolar disorder), vitamin B12 deficiency, iron deficiency anemia, patients with neurodegenerative diseases of the brain or retina or cerebrovascular diseases and those who do not agree to sign the informed consent form. Eligible patients will undergo a medical consultation, which will consist of anamnesis and physical examination and will wear a flash glucose monitor, model Freestyle Libre by Abbott, which should be used for a period of 7 to 14 days. They will complete the Three Factor Eating Questionnaire R21 (TFEQ-R21), International Physical Activity Questionnaire (IPAQ), Gold Questionnaire, Edinburgh Hypoglycemia Symptom Scale (EHSS), Rey Auditory Verbal Learning Test (RAVLT), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Trail Making Test (TMT) and Stroop Test. Will be evaluated as possible predictive factors the time elapsed from surgery, surgical technique, excess weight loss, rate of weight regain, previous diabetes mellitus, age, sex, resting heart rate, history of cholecystectomy, laboratory values of glycated hemoglobin, fasting glycemia, lipidogram and renal, thyroid and hepatic functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to GRYR and SG, for at least one year, undergoing medical follow-up at the Multiuser Clinical Research Center (CePeM) of the Pedro Ernesto University Hospital (HUPE).

Exclusion Criteria:

* patients using hypoglycemic drugs (biguanides, sulfonylureas, glinides, acarbose, GLP-1 analogues, SGLT-2 inhibitors, DPP-IV inhibitors and insulin) and hyperglycemic drugs (corticosteroids, high-dose thiazide diuretics, beta-blockers, diazoxide and octreotide) , very restrictive diets (intermittent fasting or ketogenic diet), pregnant women, kidney, heart and/or liver failure, history of neurological disorder, visual or hearing impairment, being treated for alcohol or drug abuse, severe psychiatric disorders (schizophrenia, bipolar disorder ), vitamin B12 deficiency, iron deficiency anemia, patients with neurodegenerative diseases of the brain or retina or cerebrovascular diseases and those who do not agree to sign the informed consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients submitted to GRYR and SG, for at least one year and control subjects not submitted to bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
High glucose variability | 14 days
  Interstitial blood glucose
Unawareness hypoglycemia | 14 days
  Interstitial blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Clinical and Experimental Research on Vascular Biology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided